CLINICAL TRIAL: NCT06031467
Title: Evaluation of the Effect of Erbium, Chromium:Yttrium-scandium-gallium-garnet (Er,Cr:YSGG) Laser Application on Peri-Implant Crevicular Fluid RANKL and OPG Levels in the Treatment of Peri-implantitis: A Randomized Clinical Trial
Brief Title: Er,Cr:YSGG Laser Application in Peri-implantitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Nazli Zeynep Alpaslan, DDS, PhD, Assoc. Prof. Dr, Yuzuncu Yil University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 29.01.2020/11
Record Dates: First submitted 2023-09-04; First posted 2023-09-11 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Peri-Implantitis
Keywords: Er:Cr:YSGG; biomarkers; laser; osteoprotegerin; peri-implantitis; RANKL
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-surgical mechanical therapy (Active Comparator): Titanium curettes were used for non-surgical mechanical therapy in both groups under local anesthesia. The curette was gently inserted into the peri-implant pocket and the mechanical therapy was completed with threads felt. The control group received mechanical therapy alone.
  Interventions: Device: Non-surgical mechanical therapy
- Er, Cr: YSGG laser-assisted non-surgical mechanical therapy (Active Comparator): Titanium curettes were used for non-surgical mechanical therapy in both groups under local anesthesia. The curette was gently inserted into the peri-implant pocket and the mechanical therapy was completed with threads felt. The laser group received mechanical therapy followed by Er;Cr;YSGG laser.
  Interventions: Device: Er, Cr: YSGG laser-assisted non-surgical mechanical therapy

INTERVENTIONS:
Device: Er, Cr: YSGG laser-assisted non-surgical mechanical therapy — The laser group received mechanical therapy followed by Er;Cr;YSGG laser. Laser application was performed using the bottom-up technique. Therefore, the tip was retracted about 1 mm after it was placed on the bottom of the pocket and slowly moved in the coronal direction to the parallel to the implant surface.
  Arms: Er, Cr: YSGG laser-assisted non-surgical mechanical therapy
Device: Non-surgical mechanical therapy — Traditional non surgical mechanical therapy Mechanical instrumentation in all groups was made with titanium curettes.The curette was gently inserted into the peri-implant pocket and the mechanical therapy was completed with threads felt.
  Arms: Non-surgical mechanical therapy

SUMMARY:
In the present study, investigators, aimed to evaluate the effect of erbium, chromium:yttrium-scandium-gallium-garnet (Er,Cr:YSGG) laser application combined with mechanical debridement (MD) on clinical parameters and biochemical parameters such as receptor activator of nuclear factor-kappa B ligand (RANKL) and osteoprotegerin (OPG) in patients with peri-implant diseases.

DETAILED DESCRIPTION:
Peri-implantitis is a plaque-associated which involves the tissues around dental implants characterized by inflammation and progressive loss of the supporting alveolar bone. According to a meta-analysis and systematic review, the prevalence of peri-implantitis is about 22%. Biofilm, poor plaque control, and poor dental care after dental implant are implicated in the etiology of disease.

Surface decontamination of the implant is the cornerstone of peri-implantitis treatment. However, there is no sufficient evidence to demonstrate the superiority of a specific decontamination protocol in the literature. Nevertheless, a review recommended the potential use of laser-assisted procedures as an adjunct to mechanical instrumentation and implant detoxification in both non-surgical and regenerative interventions for the treatment of peri-implant diseases. Several studies have examined the role of a variety of laser types in both periodontal and peri-implant treatments and laser application has been shown to play a central role in wound healing and tissue regeneration.

Erbium lasers such as erbium, chromium:yttrium-scandium-gallium-garnet (Er,Cr:YSGG) use mid-infrared wavelengths which are highly absorbed by water and hydroxyapatite crystals and minerals. In a recent in vitro study, Er,Cr:YSGG laser has been shown to be a safe method in the treatment of peri-implantitis with the dual wavelength protocol. In the literature, there is a limited number of studies using Er,Cr:YSGG laser in the treatment of peri-implantitis in the in vivo setting. Although limited, favorable results have been described in a case report with 18-month follow-up, case reports of including 11 patients, and randomized-controlled clinical studies. Taken together, Er,Cr:YSGG laser seems to be an effective treatment modality in reducing clinical symptoms of peri-implantitis.

The detection of specific biomarkers in the peri-implant crevicular fluid (PICF) is promising to objectively evaluate peri-implant inflammation at baseline and assess treatment efficacy. Biomarkers are host response molecules which reflect a biological state and help to distinguish healthy from diseased tissues or to evaluate disease and its severity.

Recent discoveries regarding the receptor activator of nuclear factor-kappa B ligand (RANKL) and osteoprotegerin (OPG) receptor activator that induce and inhibit osteoclast differentiation have shown that both markers play a role in the molecular network of peri-implant bone resorption. The RANKL is a member of tumor necrosis factor (TNF) superfamily which interacts on osteoclastogenesis. It is secreted by osteoblasts, fibroblasts, and activated T cells and is associated with RANK as a surface-bound molecule which stimulates osteoclast activity. On the other hand, OPG is a soluble decoy receptor for RANKL and expressed by osteoblasts. It also inhibits the osteoclast differentiation and prevents the interaction between RANKL and RANK.

Previous studies have shown high RANKL levels in the crevicular fluid of patients with periodontitis and peri-implantitis compared to healthy dental sites. However, there are controversial results regarding OPG. Several studies have reported significantly higher OPG and RANK levels at peri-implant disease sites compared to healthy implant sites. In addition, significantly higher RANKL protein levels and significantly lower OPG protein levels have been reported in periodontitis tissue. In a study, the PICF level of soluble RANKL was not significantly correlated with clinical parameters and OPG. However, the authors found a positive correlation between the total OPG level and PICF volume, bleeding on probing (BoP) and gingival index (GI).

To the best of investigators' knowledge, there is no study investigating the effect of Er,Cr:YSGG laser as an adjunct to mechanical debridement (MD) on RANKL and OPG in the treatment of peri-implantitis. In the present study, investigators, therefore aimed to evaluate the effect of Er,Cr:YSGG laser application combined with MD on clinical parameters and biochemical parameters such as RANKL and OPG in patients with peri-implant diseases.

ELIGIBILITY:
Inclusion Criteria:

* bone loss as evidenced by X-ray and inflammatory symptoms in the soft tissue, bleeding and/or suppuration around the implant compatible with peri-implantitis (each patient had a single dental implant or the implant in the deepest pathological pocket not requiring surgical intervention was chosen in case of peri-implantitis in multiple implants);
* radiotherapy or chemotherapy-naïve patients;
* having no bone disease such as osteoporosis or osteopetrosis;
* receiving no bisphosphonate therapy;
* having functional prosthetic loading on the implant for at least six months
* requiring no advanced surgical technique for the treatment of peri-implantitis.

Exclusion Criteria:

* having systemic diseases such as diabetes, autoimmune disorder, renal or hepatic impairment;
* having uncontrolled periodontal disease in natural teeth existing in the mouth;
* smoking habit;
* having parafunctional habits which affect osseointegration of the dental implant;
* receiving antibiotherapy three months before the diagnosis of peri-implantitis;
* having non-osseointegrated dental implant;
* pregnancy and lactation.

Ages: 28 Years to 63 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2022-04-08 (Actual); Study Completion 2022-04-08 (Actual)

PRIMARY OUTCOMES:
Probing depth (mm) | 6 months
  Probing depth (PD) (distance from peri-implant margin to peri-implant pocket base) was measured with a plastic probe in 4 regions (mesial, buccal, distal, lingual / palatial) of each implant and recorded as mm.
Receptor activator of nuclear factor-kappa B ligand (RANKL) level (pg/mL) | 6 months
  All PICF samples were collected before clinical measurements. During sample collection, the implants were isolated using cotton rolls and dried gently with an air freshener, and paper strips were advanced into the pocket until resistance was felt. The paper strips were kept in the peri-implant pocket for 30 sec. Paper strips were placed in 500-µL sterilized Eppendorf® tubes to which phosphate-buffered saline (PBS) was added. All samples were kept at -40° until analysis. The enzyme-linked immunosorbent assay (ELISA) was used to measure RANKL levels in the PICF samples in accordance with the manufacturer's instructions.
Osteoprotegerin (OPG) level (ng/mL) | 6 months
  All PICF samples were collected before clinical measurements. During sample collection, the implants were isolated using cotton rolls and dried gently with an air freshener, and paper strips were advanced into the pocket until resistance was felt. The paper strips were kept in the peri-implant pocket for 30 sec. Paper strips were placed in 500-µL sterilized Eppendorf® tubes to which phosphate-buffered saline (PBS) was added. All samples were kept at -40° until analysis. The enzyme-linked immunosorbent assay (ELISA) was used to measure OPG levels in the PICF samples in accordance with the manufacturer's instructions.

SECONDARY OUTCOMES:
Plaque index score (0-3) | 6 months
  Plaque index was measured from the 4 surfaces of each implant. The plaque index score of each implant was calculated with Silness-Loe plaque index by dividing the total value by 4.
  0:absence of microbial plaque
  1. Thin film of microbial plaque along the free peri-implant margin
  2. moderate accumulation with plaque in the sulcus
  3. large amount of plaque in sulcus or pocket along the free peri-implant margin
Gingival index score (0-3) | 6 months
  The gingival index was measured from the 4 surfaces of each implant. The gingival index score of each implant was calculated with Silness-Loe gingival index by dividing the total value by 4.
  0:Normal gingiva
  1. Mild inflammation: slight change in color, slight oedema, no bleeding on probing
  2. Moderate inflammation: redness,oedema and glazing, bleeding on probing
  3. Severe inflammation: marked redness and oedema, ulceration, tendency to spontaneous bleeding
Bleeding on probing (percentage) | 6 months
  Bleeding on probing was measured from 4 surfaces of each implant. If there is bleeding after probing, it is recorded as +, if there is no bleeding it is recorded as _. Gingival bleeding index is calculated as a percentage of affected sites.

CONTACTS AND LOCATIONS:
Overall Officials: Nazli Zeynep Alpaslan, PhD, Principal Investigator — Yuzuncu Yil University; Dicle Altindal, PhD, Study Chair — Yuzuncu Yil University; Damla Akbal, PhD, Study Chair — Private Dental Clinic; Ahmet Cemil Talmac, PhD, Study Chair — Yuzuncu Yil University; Serap Keskin Tunc, PhD, Study Chair — Saglik Bilimleri Universitesi; Abdullah Seckin Ertugrul, PhD, Study Chair — Izmir Katip Celebi University
Locations (1):
- Nazli Zeynep Alpaslan, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Alpaslan Yayli NZ, Talmac AC, Keskin Tunc S, Akbal D, Altindal D, Ertugrul AS. Erbium, chromium-doped: yttrium, scandium, gallium, garnet and diode lasers in the treatment of peri-implantitis: clinical and biochemical outcomes in a randomized-controlled clinical trial. Lasers Med Sci. 2022 Feb;37(1):665-674. doi: 10.1007/s10103-021-03436-5. Epub 2021 Oct 12. PMID 34637055